CLINICAL TRIAL: NCT03404518
Title: Quantifying Narcotic Use in Outpatient Otolaryngology Procedures
Brief Title: Patient Narcotic Requirements After Outpatient Otolaryngology Procedures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Jared Inman, Associate Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5170252
Record Dates: First submitted 2018-01-11; First posted 2018-01-19 (Actual); Results first posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-02

CONDITIONS: Outpatient Surgery; Pain, Postoperative
Keywords: Thyroidectomy; Parotidectomy; Tympanoplasty; Mastoidectomy; Septoplasty; Sinus Surgery; Postoperative pain; Outpatient surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — oxycodone-acetaminophen; Narcotics; Ibuprofen; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of two groups prior to surgery. All patients will be prescribed both Hydrocodone/acetaminophen and Ibuprofen. Group 1 will take the narcotic medication for initial pain control followed by Ibuprofen if pain is not adequately controlled. Group 2 will take Ibuprofen for initial pain control followed by the narcotic medication if pain is not adequately controlled.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Norco and Ibuprofen (Experimental): This group will take Hydrocodone/acetaminophen 5mg/325mg every 6 hours as needed for pain control as first line intervention.
  If pain is not controlled after 60 minutes then can take Ibuprofen 600mg every 6 hours as needed for additional pain control.
  Interventions: Drug: Norco
- Ibuprofen and Norco (Active Comparator): This group will take Ibuprofen 600mg every 6 hours as needed for pain control as first line intervention.
  If pain is not controlled after 60 minutes then can take Hydrocodone/acetaminophen 5mg/325mg every 6 hours as needed for additional pain control.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Norco — Hydrocodone/Acetaminophen as first line therapy every 6 hours as needed for pain control
  Other Names: Hydrocodone/Acetaminophen; Narcotic
  Arms: Norco and Ibuprofen
Drug: Ibuprofen — Ibuprofen as first line therapy every 6 hours as needed for pain control
  Other Names: NSAID; Motrin; Advil
  Arms: Ibuprofen and Norco

SUMMARY:
Patient's pain level and narcotic requirements will be evaluated after routine outpatient Otolaryngology procedures. This will be done by having study participants record their pain level and medication usage from home.

DETAILED DESCRIPTION:
It is routine practice to give narcotic medication after surgery for pain control however the abuse of prescription medications has become the fastest growing drug problem in the United States. Research has shown that post operative pain for some common Ear, Nose, and Throat (ENT) procedures are not severe but there is limited data looking at patient narcotic needs and their usage pattern to help inform physicians on how much to prescribe.

The objective of this study is to evaluate patient pain level in the immediate post-operative period and quantify pain medication usage in patients who undergo outpatient ENT surgeries.

Patients who undergo the following procedures will be invited to participate: thyroidectomy, parathyroidectomy, parotidectomy, tympanoplasty, mastoidectomy, endoscopic sinus surgery, and septoplasty. All patients will receive Hydrocodone/acetaminophen and Ibuprofen in standard dosage and assigned to one of two groups before surgery. Group 1 will use the narcotic medication for pain control and ibuprofen for breakthrough pain. Group 2 will use ibuprofen for pain control and the narcotic medication for breakthrough. Patients will fill out a data sheet for 7 days recording their pain level three times per day as well as pain medication usage for each day. This will be collected on their first clinic visit after surgery at which point the patient's involvement is completed.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing one of the following outpatient procedure:

* Septoplasty
* Unilateral or Bilateral Functional endoscopic sinus surgery
* Tympanomastoidectomy
* Tympanoplasty
* Total or Partial Thyroidectomy
* Parathyroidectomy
* Parotidectomy.
* Age >18 years and < 89 years

Exclusion Criteria:

* Age < 18 years or > 89 years
* Post operative hospital admission
* Allergy to Hydrocodone
* Allergy or contraindication to Ibuprofen or NSAIDs
* Pregnancy
* Hepatic disease
* Chronic kidney disease
* Sickle cell anemia

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Inman, MD, Principal Investigator — Loma Linda University Health System
Locations (2):
- United States (2):
  - Loma Linda University Medical Center, Loma Linda, California
  - Loma Linda University Surgical Hospital, Loma Linda, California

IPD SHARING:
Plan to Share IPD: No
Collected data will be analyzed and published. Meaningful data will be available through published material.

REFERENCES:
- [Background] Sommer M, Geurts JW, Stessel B, Kessels AG, Peters ML, Patijn J, van Kleef M, Kremer B, Marcus MA. Prevalence and predictors of postoperative pain after ear, nose, and throat surgery. Arch Otolaryngol Head Neck Surg. 2009 Feb;135(2):124-30. doi: 10.1001/archoto.2009.3. PMID 19221238
- [Background] Foghsgaard S, Foghsgaard J, Homoe P. Early post-operative morbidity after superficial parotidectomy: a prospective study concerning pain and resumption of normal activity. Clin Otolaryngol. 2007 Feb;32(1):54-7. doi: 10.1111/j.1365-2273.2007.01315.x. PMID 17298314
- [Background] Song CM, Ji YB, Bang HS, Kim KR, Kim H, Tae K. Postoperative Pain After Robotic Thyroidectomy by a Gasless Unilateral Axillo-Breast or Axillary Approach. Surg Laparosc Endosc Percutan Tech. 2015 Dec;25(6):478-82. doi: 10.1097/SLE.0000000000000204. PMID 26422088
- [Background] van Dijk JF, Kappen TH, Schuurmans MJ, van Wijck AJ. The Relation Between Patients' NRS Pain Scores and Their Desire for Additional Opioids after Surgery. Pain Pract. 2015 Sep;15(7):604-9. doi: 10.1111/papr.12217. Epub 2014 Apr 16. PMID 24735082
- [Background] van Dijk JF, van Wijck AJ, Kappen TH, Peelen LM, Kalkman CJ, Schuurmans MJ. Postoperative pain assessment based on numeric ratings is not the same for patients and professionals: a cross-sectional study. Int J Nurs Stud. 2012 Jan;49(1):65-71. doi: 10.1016/j.ijnurstu.2011.07.009. Epub 2011 Aug 15. PMID 21840522
- [Background] Gerbershagen HJ, Rothaug J, Kalkman CJ, Meissner W. Determination of moderate-to-severe postoperative pain on the numeric rating scale: a cut-off point analysis applying four different methods. Br J Anaesth. 2011 Oct;107(4):619-26. doi: 10.1093/bja/aer195. Epub 2011 Jun 30. PMID 21724620
- [Background] Ossiander EM. Using textual cause-of-death data to study drug poisoning deaths. Am J Epidemiol. 2014 Apr 1;179(7):884-94. doi: 10.1093/aje/kwt333. Epub 2014 Feb 11. PMID 24521559
- See also: CDC report on opioid related deaths — https://www.cdc.gov/mmwr/volumes/65/wr/mm655051e1.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Norco and Ibuprofen: This group will take Hydrocodone/acetaminophen 5mg/325mg every 6 hours as needed for pain control as first line intervention.
  If pain is not controlled after 60 minutes then can take Ibuprofen 600mg every 6 hours as needed for additional pain control.
  Norco: Hydrocodone/Acetaminophen as first line therapy every 6 hours as needed for pain control
- Ibuprofen and Norco: This group will take Ibuprofen 600mg every 6 hours as needed for pain control as first line intervention.
  If pain is not controlled after 60 minutes then can take Hydrocodone/acetaminophen 5mg/325mg every 6 hours as needed for additional pain control.
  Ibuprofen: Ibuprofen as first line therapy every 6 hours as needed for pain control
Period: Overall Study
Arm/Group | Norco and Ibuprofen | Ibuprofen and Norco
Started | 97 | 88
Completed | 56 | 52
Not Completed | 41 | 36
Not completed — Lost to Follow-up | 28 | 30
Not completed — Protocol Violation | 13 | 6

BASELINE CHARACTERISTICS:
Population: Patients who completed and returned pain data entry
Groups:
- Total: Total of all reporting groups
Arm/Group | Norco and Ibuprofen | Ibuprofen and Norco | Total
Number analyzed (Participants) | 56 | 52 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (17) | 52.9 (17) | 53 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 26 | 63
  Male | 19 | 26 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Prior Narcotic use [Count of Participants; unit: Participants] | 4 | 3 | 7
Chronic Pain [Count of Participants; unit: Participants] | 15 | 11 | 26
Surgery Length [Mean (Standard Deviation); unit: minutes] | 94.4 (43) | 95.3 (43) | 94.8 (42.7)
Revision Surgery [Count of Participants; unit: Participants] | 19 | 16 | 35

OUTCOME MEASURES:

1. Primary Outcome: Narcotic Usage
Description: The average number of narcotic pills needed or used for pain control
Time Frame: First 7 days after surgery
Measure: Mean (95% Confidence Interval); unit: Pills
Arm/Group | Norco and Ibuprofen | Ibuprofen and Norco
Number analyzed (Participants) | 56 | 52
Pills | 4.9 [3.6 to 6.3] | 2.0 [0.9 to 3.1]

2. Secondary Outcome: Patient Pain Level
Description: The average reported pain score using the Numeric Rating Scale (0-10) with 0 representing no pain and 10 as worse imaginable pain.
Time Frame: Average reported pain for first 7 days after surgery
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Norco and Ibuprofen | Ibuprofen and Norco
Number analyzed (Participants) | 56 | 52
Scores on a scale | 3.5 [2.8 to 4.1] | 2.8 [2.2 to 3.4]

3. Secondary Outcome: Ibuprofen Usage
Description: The average number of ibuprofen pills needed or used for pain control
Time Frame: First 7 days after surgery
Measure: Mean (95% Confidence Interval); unit: pills
Arm/Group | Norco and Ibuprofen | Ibuprofen and Norco
Number analyzed (Participants) | 56 | 52
pills | 4.5 [3.2 to 5.7] | 7.7 [5.8 to 9.6]

ADVERSE EVENTS:
Time Frame: Days 1-7 following surgery or until the first follow up appointment with provider up to 14 days following surgery
Description: Adverse event would include any report or contact with the clinic to request for additional medication refills, emergency room visit related to the surgery, any additional procedure necessary due to complications from the surgery
Arm/Group | Norco and Ibuprofen | Ibuprofen and Norco
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/88
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/88
Other Adverse Events (participants affected / at risk) | 4/97 | 3/88
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Norco and Ibuprofen (N=97) | Ibuprofen and Norco (N=88)
Headache (Nervous system disorders) | 1 | 0 — Patient reported headache
Drainage from surgical site (Surgical and medical procedures) | 1 | 1 — Patient had additional blood tinged secretion from surgical site
Uncontrolled pain (Surgical and medical procedures) | 1 | 2 — Patient requiring additional pain medication refill
Nausea (Gastrointestinal disorders) | 1 | 0 — Patient reported nausea

LIMITATIONS AND CAVEATS:
Some patients chose to not follow study instructions strictly and utilized ibuprofen therapy as primary analgesic treatment instead of their opioid medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT03404518/Prot_SAP_001.pdf